CLINICAL TRIAL: NCT05269940
Title: A Phase I/II Study Evaluating ZX-101A in Patients with Relapsed/Refractory Hematological Malignancies
Brief Title: A Study to Evaluate Activity, Safety and Tolerability of ZX-101A in Relapsed/Refractory Hematological Malignancies
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nanjing Zenshine Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ZX-101A-202
Record Dates: First submitted 2022-01-23; First posted 2022-03-08 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Non Hodgkin Lymphoma; Peripheral T Cell Lymphoma; CLL/SLL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Lymphoma, T-Cell, Peripheral

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- ZX-101A Dose Level A (Experimental): ZX-101A administered orally at level A once daily
  Interventions: Drug: ZX-101A
- ZX-101A Dose Level B (Experimental): ZX-101A administered orally at level B once daily
  Interventions: Drug: ZX-101A
- ZX-101A Dose Level C (Experimental): ZX-101A administered orally at level C once daily
  Interventions: Drug: ZX-101A
- ZX-101A Dose Level D (Experimental): ZX-101A administered orally at level D once daily
  Interventions: Drug: ZX-101A
- ZX-101A Dose Level E (Experimental): ZX-101A administered orally at level E once daily
  Interventions: Drug: ZX-101A

INTERVENTIONS:
Drug: ZX-101A — oral dosing, once daily

SUMMARY:
ZX-101A-202 is a Phase I, open-label, multicenter study, a single-agent dose-escalation and dose-expansion study of ZX-101A. It is designed to evaluate the safety, tolerability, pharmacokinetics, pharmacokinetics, efficacy and antitumor activity of ZX-101A in patients with relapsed/refractory hematological malignancies.

DETAILED DESCRIPTION:
Phase I includes two parts: dose escalation and dose expansion. It's mainly to explore the safety and tolerability of ZX-101A in patients with relapsed/ refractory hematological malignancies [Chronic Lymphocytic Leukemia (CLL)/ Small Lymphocytic Lymphoma (SLL), indolent NHL, and other NHL subtypes], and to determine RP2D.

* Part 1. ZX-101A dose escalation
* Part 2. ZX-101A dose expansion in two specific types of lymphoma, i.e. PTCL /CTCL or one B-iNHL.

ELIGIBILITY:
Inclusion Criteria:

* Males and females who are ≥ 18 years old
* Minimum life expectancy ≥ 3 months (determined by investigator assessment)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to1.
* Histopathological and cytological confirmed diagnosis of hematological malignancies.
* Phase I dose expansion and phase II studies require at least 1 measurable lesion, including cutaneous T-cell lymphoma [CTCL] without evidence of skin involvement.
* Acceptable bone marrow function.
* Acceptable organ function: creatinine clearance ≥ 60 mL/min calculated according to institutional standard practice assessment (according to the Cockcroft-Gault formula) for kidney function; AST and ALT ≤ 2.5 x upper limit of normal (ULN) (AST and ALT ≤ 4 x ULN in subjects with liver involvement); total bilirubin ≤ 1.5 x ULN (total bilirubin ≤ 3 in subjects with Gilbert syndrome ×ULN) for liver function.
* No transfusion or cytokine support for ≥ 2 weeks before first dosing.
* Ability to swallow oral medication.
* Negative serum pregnancy test in women of childbearing potential at screening.
* Females of childbearing potential and males with female partners of childbearing potential must agree to use effective contraception during the study period and for 6 months (females) or 3 months (males) after the last dose of ZX-101A.
* Men must agree to no sperm donation during the study and for 3 months after the last dose of ZX-101A.
* Understands the requirements of the study, is willing to comply with all study procedures and signed the IRB-approved informed consent.

Exclusion Criteria:

* Previous use of PI3K δ/γ dual inhibitors
* Received approved anti-cancer drugs within 28 days (42 days for nitrosoureas) or 5 half-lives, whichever is longer.
* Radiation treatment within 2 weeks prior to first dose of study treatment.
* Received investigational study drug within 28 days (or 5 half-lives, whichever is longer).
* Received organ transplantation in the past (hematopoietic stem cell transplantation in the past is allowed).
* Major surgery within 28 days prior to the first dose of study drug
* Has not recovered from adverse events from prior anti-cancer treatment (with exception of alopecia).
* Concurrent participation in another therapeutic treatment trial.
* Those who have been vaccinated with live vaccines or live attenuated vaccines within 30 days before the first administration, and seasonal influenza vaccines without live viruses are allowed.
* Received warfarin or factor Xa inhibitor within 5 half-lives before the first dose of study drug.
* With central nervous system (CNS) involvement or active leptomeningeal disease.
* History of other malignancy within the past 5 years, unless cured by surgery and sustained disease-free survival.
* CLL with Richter transformation.
* Active autoimmune hemolytic anemia (AIHA) or idiopathic thrombocytopenic purpura (ITP)
* Chronic immunosuppression conditions.
* QTcF interval > 480 msec; echocardiographic detection of left ventricular ejection fraction < 45%.
* Uncontrolled systemic diseases, including myocardial infarction or bypass, stent surgery, or other heart disease, in the judgement of the investigator, inappropriate for enrollment.
* Active uncontrolled infection within 14 days before first dosing.
* Active infection of Hepatitis B virus or hepatitis C virus; history of HIV infection.
* History of drug-induced liver injury, chronic active hepatitis, alcoholic liver disease, nonalcoholic steatohepatitis, primary biliary cirrhosis, persistent extrahepatic obstruction due to gallstones, cirrhosis or portal vein history of hypertension.
* History of interstitial lung disease, hypersensitivity pneumonitis, pulmonary fibrosis, radiation pneumonitis and severe pulmonary function impairment, or other pulmonary diseases that significantly affect the safety or compliance of patients after being evaluated and included by the investigator.
* Gastrointestinal dysfunction, including motility or malabsorption syndromes or inflammatory bowel disease which could limit absorption of study drug.
* Any concurrent uncontrolled illness, including mental illness or substance abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2022-02-17 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2024-07-05 (Actual)

PRIMARY OUTCOMES:
Defining the RP2D of ZX-101A | From Day 1 of Cycle 1 (each cycle is 28 days) until 28 days after the last dose (up to 2 years)
  To assess number of patients experiencing dose-limiting toxicities (DLTs)
To examine the incidence of clinical and laboratory adverse events after multiple doses of ZX-101A | From Day 1 of Cycle 1 (each cycle is 28 days) until 28 days after the last dose (up to 2 years)
  Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability]

SECONDARY OUTCOMES:
Objective response rate (ORR) | Up to 2 years
  To evaluate the objective response rate (ORR) as determined by the specific disease response criteria
Duration of response (DoR) | Up to 2 years
  To examine the duration of response (DoR), defined as time from the date of first documentation of response to the date of the first documentation of progressive disease (PD), or death due to any cause
Progression free survival (PFS) | Up to 2 years
  To examine the the progression free survival (PFS), defined as time from the date of first dose of study treatment to the first date of documentation of PD, or death due to any cause
Overall survival (OS) | Up to 2 years
  To examine the overall survival (OS), defined as time from the date of first dose of study treatment to death due to any cause
Plasma Concentration of ZX-101A | Cycle1Day1 pre-dose and post-dose 0.5, 1 , 2, 4, 6, 8, 24, 48, 72, 96 hours; Cycle1Day13, Day14, Day15 pre-dose and post-dose 0.5, 1, 2, 4 , 6, 8 and 24 hours; Cycle2Day1 pre-dose. Each cycle is 28 days.
  To assess the pharmacokinetic (PK) characteristics of ZX-101A and its major metabolites (if applicable) in part 1
Phospho-AKT (p-AKT) levels in whole blood | Cycle1Day1 pre-dose and post-dose 1 hour and 24 hours. Each Cycle is 28 days.
  To evaluate the differences phospho-AKT (p-AKT) levels in whole blood before and after single oral dose of ZX-101A.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaolin Qin, PhD, Study Director — Zenshine Pharmaceutical, Inc.
Locations (3):
- China (3):
  - Anhui Medical University No.4 Affiliated Hospital, Hefei, Anhui
  - Wuhan Union Hospital, Wuhan, Hubei
  - Hunan Tumor Hospital, Changsha, Hunan